CLINICAL TRIAL: NCT02911584
Title: Laparoscopic Sacrocolpopexy Versus POPS in the Surgical Management of Pelvic Organ Prolapse: A Prospective Randomized Trial
Brief Title: Laparoscopic Sacrocolpopexy Versus POPS in the Management of Pelvic Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Miulli General Hospital (Other)
Responsible Party: Principal Investigator, Valeria Tagliaferri, Medical Doctor, Miulli General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP1
Record Dates: First submitted 2016-09-15; First posted 2016-09-22 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Sacral colpopexy (Active Comparator): Laparoscopic procedure
  Interventions: Procedure: Laparoscopic procedure
- POPS (Active Comparator): Laparoscopic procedure: Pelvic Organs Prolapse Suspension
  Interventions: Procedure: Laparoscopic procedure

INTERVENTIONS:
Procedure: Laparoscopic procedure

SUMMARY:
This is the first study comparing the laparoscopic sacropexy with Pelvic Organs Prolapse Suspension (POPS) to treat pelvic organ prolapse. This prospective randomized surgical trial is designed to test the clinical and functional effects of the two different laparoscopic procedures in terms of anatomical correction of the prolapse, post-operative and long term morbidity, rate of recurrence and subjective satisfaction of the patient evaluated by a quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who required surgical treatment for symptomatic pelvic organ prolapse stage ≥ 2 with or without stress urinary incontinence

Exclusion Criteria:

* Age > 70 years
* Severe cardiovascular or respiratory disease
* Pregnancy
* Previous surgical procedure for POP correction

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10; Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with anatomical correction of the prolapse | up to 6 months
  Anatomical correction of the prolapse evaluated by gynecological visit

SECONDARY OUTCOMES:
Rate of recurrence | up to 6 months
Post operative quality of life | up to 6 months
  Subjective satisfaction of the patient evaluated by a quality of life questionnaire.